CLINICAL TRIAL: NCT06335160
Title: Clinical Study to Evaluate the Possible Efficacy and Safety of Mebendazole in Patients With Ulcerative Colitis Treated With Mesalamine
Brief Title: Possible Efficacy and Safety of Mebendazole in Patients With Ulcerative Colitis Treated With Mesalamine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Eman Elberri, Lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mebendazole Ulcerative Colitis
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Ulcerative Colitis
Keywords: MBZ, UC
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mebendazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): control group (Mesalamine group, n =23) who will receive 1 g mesalamine three times daily for 6 months.
- Treatment Group (Active Comparator): Treatment group( mebendazole group, n = 23) which will receive the standard treatment for UC plus mebendazole 500 mg twice daily for 6 months
  Interventions: Drug: Mebendazole

INTERVENTIONS:
Drug: Mebendazole — mebendazole group, n = 23) which will receive the standard treatment for UC plus mebendazole 500 mg twice daily for 6 months
  Arms: Treatment Group

SUMMARY:
To evaluate the possible efficacy and safety of mebendazole in patients with ulcerative colitis treated with mesalamine

DETAILED DESCRIPTION:
A randomized, controlled, and parallel study will comprise 46 patients with UC. Patients will be recruited from GastroEnterology Department, Mansoura University Hospital.

The participants will be randomly assigned into two groups as follow:

Group 1: control group (Mesalamine group, n =23) who will receive 1 g mesalamine three times daily for 6 months.

Group 2: (mebendazole group, n = 23) which will receive the standard treatment for UC plus mebendazole 500 mg twice daily for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old Both male and female will be included Mild and moderate UC patients diagnosed and confirmed by endoscope Patient treated with 5-aminosalislic acid (mesalamine)

Exclusion Criteria:

* - Patients with severe UC
* Significant liver and kidney function abnormalities
* Diabetic patients
* Patients with Colorectal cancer patients
* Patients taking rectal or systemic steroids
* Patients on immunosuppressants or biological therapies
* Addiction to alcohol and / or drugs
* Known allergy to the studied medications
* History of complete or partial colectomy.
* Patients with congestive heart failure, other heart disease (arrhythmia, ischemic heart disease including angina and myocardial infarction).
* Patients with other inflammatory diseases and active infection.
* Patients with stressful condition (COPD, morbid obesity).
* Patients with liver disease.
* Patients with thrombocytopenia and neutropenia.
* Patients with any type of seizures (case report for mebendazole induced convulsion).
* Patients with renal disease (case report for mebendazole induced nephrotoxicity).
* Patients with coagulation disorders.
* Patients on metronidazole (to avoid Stevens-Johnson syndrome).
* Patients with hypersensitivity to mebendazole, albendazole or benzimidazole
* Patients using antioxidants.
* Pregnant and lactating females.
* Patients receiving, metronidazole, warfarin, low dose of aspirin, clopidogril, enzyme inducers (phenytoin, carbamazepine) and inhibitors (valoproate) to avoid potential pharmacodynamics and pharmacokinetic interactions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
change in disease activity | change in baseline
  Disease severity which will be assessed according to the modified Truelove and Witt's classification based on number of bloody stools per day plus one or more of 4 additional criteria including pulse, temperature, hemoglobin and Erythrocyte sedimentation rate (ESR) . Remission will be defined as disappearance or improvement of symptoms such as normal stool and stooling pattern without blood, no fever, no tachycardia, hemoglobin level normal or returning toward normal, ESR normal or returning toward normal, and patient gaining weight.
change in Partial Mayo Scoring Index (PMSI) assessment for Ulcerative Colitis Activity | change in baseline
  depends on three items; stool frequency, rectal bleeding (blood in stool) and Physician's Global Assessment. Each item has a score from 0 to 3 and total PMSI is the sum of scores for the three items.
  Remission is defined as total PMSI = 0-1, mild disease is defined as total PMSI = 2-4, moderate disease is defined as total PMSI = 5-6 and severe disease is defined as total PMSI =7-9.

SECONDARY OUTCOMES:
Change in Hemoglobin Concentration | Blood samples will be taken from all patients at baseline then six months of therapy
  Enzyme-linked immunosorbent assay (ELISA)
Change in Erythrocyte sedimentation rate (ESR) | Blood samples will be taken from all patients at baseline then six months of therapy
  Enzyme-linked immunosorbent assay (ELISA)
Change in Serum albumin | Blood samples will be taken from all patients at baseline then six months of therapy
  Enzyme-linked immunosorbent assay (ELISA)
Change in Serum Interleukin -6 (IL-6) | Blood samples will be taken from all patients at baseline then six months of therapy
  Enzyme-linked immunosorbent assay (ELISA)
Change in Serum Nitric oxide (NO) | Blood samples will be taken from all patients at baseline then six months of therapy
  Enzyme-linked immunosorbent assay (ELISA)
Change in Serum Intra cellular adhesion molecule 1 (ICAM-1) | Blood samples will be taken from all patients at baseline then six months of therapy
  Enzyme-linked immunosorbent assay (ELISA)

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta Unuversity, Tanta, Egypt

REFERENCES:
- [Background] Andersson CR, Selvin T, Blom K, Rubin J, Berglund M, Jarvius M, Lenhammar L, Parrow V, Loskog A, Fryknas M, Nygren P, Larsson R. Mebendazole is unique among tubulin-active drugs in activating the MEK-ERK pathway. Sci Rep. 2020 Aug 4;10(1):13124. doi: 10.1038/s41598-020-68986-0. PMID 32753665
- [Background] Elayapillai S, Ramraj S, Benbrook DM, Bieniasz M, Wang L, Pathuri G, Isingizwe ZR, Kennedy AL, Zhao YD, Lightfoot S, Hunsucker LA, Gunderson CC. Potential and mechanism of mebendazole for treatment and maintenance of ovarian cancer. Gynecol Oncol. 2021 Jan;160(1):302-311. doi: 10.1016/j.ygyno.2020.10.010. Epub 2020 Oct 31. PMID 33131904
- [Background] Eskandari M, Asgharzadeh F, Askarnia-Faal MM, Naimi H, Avan A, Ahadi M, Vossoughinia H, Gharib M, Soleimani A, Naghibzadeh N, Ferns G, Ryzhikov M, Khazaei M, Hassanian SM. Mebendazole, an anti-helminth drug, suppresses inflammation, oxidative stress and injury in a mouse model of ulcerative colitis. Sci Rep. 2022 Jun 17;12(1):10249. doi: 10.1038/s41598-022-14420-6. PMID 35715495
- [Background] Ford AC, Achkar JP, Khan KJ, Kane SV, Talley NJ, Marshall JK, Moayyedi P. Efficacy of 5-aminosalicylates in ulcerative colitis: systematic review and meta-analysis. Am J Gastroenterol. 2011 Apr;106(4):601-16. doi: 10.1038/ajg.2011.67. Epub 2011 Mar 15. PMID 21407188
- [Background] Guerini AE, Triggiani L, Maddalo M, Bonu ML, Frassine F, Baiguini A, Alghisi A, Tomasini D, Borghetti P, Pasinetti N, Bresciani R, Magrini SM, Buglione M. Mebendazole as a Candidate for Drug Repurposing in Oncology: An Extensive Review of Current Literature. Cancers (Basel). 2019 Aug 31;11(9):1284. doi: 10.3390/cancers11091284. PMID 31480477
- [Background] Hegazy SK, El-Azab GA, Zakaria F, Mostafa MF, El-Ghoneimy RA. Mebendazole; from an anti-parasitic drug to a promising candidate for drug repurposing in colorectal cancer. Life Sci. 2022 Jun 15;299:120536. doi: 10.1016/j.lfs.2022.120536. Epub 2022 Apr 3. PMID 35385794
- [Background] Irvine EJ, Zhou Q, Thompson AK. The Short Inflammatory Bowel Disease Questionnaire: a quality of life instrument for community physicians managing inflammatory bowel disease. CCRPT Investigators. Canadian Crohn's Relapse Prevention Trial. Am J Gastroenterol. 1996 Aug;91(8):1571-8. PMID 8759664
- [Background] Jena G, Trivedi PP, Sandala B. Oxidative stress in ulcerative colitis: an old concept but a new concern. Free Radic Res. 2012 Nov;46(11):1339-45. doi: 10.3109/10715762.2012.717692. Epub 2012 Sep 5. PMID 22856328
- [Background] Kobayashi T, Siegmund B, Le Berre C, Wei SC, Ferrante M, Shen B, Bernstein CN, Danese S, Peyrin-Biroulet L, Hibi T. Ulcerative colitis. Nat Rev Dis Primers. 2020 Sep 10;6(1):74. doi: 10.1038/s41572-020-0205-x. PMID 32913180
- [Background] Puente S, Lago M, Subirats M, Sanz-Esteban I, Arsuaga M, Vicente B, Alonso-Sardon M, Belhassen-Garcia M, Muro A. Imported Mansonella perstans infection in Spain. Infect Dis Poverty. 2020 Jul 23;9(1):105. doi: 10.1186/s40249-020-00729-9. PMID 32703283
- [Background] Sturm A, Maaser C, Calabrese E, Annese V, Fiorino G, Kucharzik T, Vavricka SR, Verstockt B, van Rheenen P, Tolan D, Taylor SA, Rimola J, Rieder F, Limdi JK, Laghi A, Krustins E, Kotze PG, Kopylov U, Katsanos K, Halligan S, Gordon H, Gonzalez Lama Y, Ellul P, Eliakim R, Castiglione F, Burisch J, Borralho Nunes P, Bettenworth D, Baumgart DC, Stoker J; European Crohn's and Colitis Organisation [ECCO] and the European Society of Gastrointestinal and Abdominal Radiology [ESGAR]. ECCO-ESGAR Guideline for Diagnostic Assessment in IBD Part 2: IBD scores and general principles and technical aspects. J Crohns Colitis. 2019 Mar 26;13(3):273-284. doi: 10.1093/ecco-jcc/jjy114. No abstract available. PMID 30137278
- [Background] Tolomeo M, Colomba C, Meli M, Cascio A. Hepatotoxicity caused by mebendazole in a patient with Gilbert's syndrome. J Clin Pharm Ther. 2019 Dec;44(6):985-987. doi: 10.1111/jcpt.13033. Epub 2019 Aug 18. PMID 31423600
- [Background] Wildenberg ME, Levin AD, Ceroni A, Guo Z, Koelink PJ, Hakvoort TBM, Westera L, Bloemendaal FM, Brandse JF, Simmons A, D'Haens GR, Ebner D, van den Brink GR. Benzimidazoles Promote Anti-TNF Mediated Induction of Regulatory Macrophages and Enhance Therapeutic Efficacy in a Murine Model. J Crohns Colitis. 2017 Dec 4;11(12):1480-1490. doi: 10.1093/ecco-jcc/jjx104. PMID 28961920
- [Background] Younis NS, Ghanim AMH, Saber S. Mebendazole augments sensitivity to sorafenib by targeting MAPK and BCL-2 signalling in n-nitrosodiethylamine-induced murine hepatocellular carcinoma. Sci Rep. 2019 Dec 13;9(1):19095. doi: 10.1038/s41598-019-55666-x. PMID 31836811
- [Background] Zingarelli B, Szabo C, Salzman AL. Reduced oxidative and nitrosative damage in murine experimental colitis in the absence of inducible nitric oxide synthase. Gut. 1999 Aug;45(2):199-209. doi: 10.1136/gut.45.2.199. PMID 10403731